CLINICAL TRIAL: NCT06898320
Title: Prediction of Cardiac Injury Due to Anthracycline Chemotherapy in Paediatric Oncological Patients Using Advanced Echocardiography and Circulating Biomarkers.
Brief Title: Cardiac Injury Due to Anthracycline in Paediatric Oncological Patients
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 44/2023
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Heart Injuries; Anthracycline
Keywords: Cardiac injury; Anthracycline chemotherapy; echocardiography; Circulating biomarkers
MeSH Terms: conditions — Heart Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anthracycline therapy: Paediatric oncological patients receiving anthracycline chemotherapy

SUMMARY:
The study investigates the role of echocardiography and of serum biomarkers (NT-proBNP, cardiac Troponin-I) in predicting cardiac injury in a cohort of paediatric oncological patients treated with Anthracycline chemotherapy.

DETAILED DESCRIPTION:
Anthracycline chemotherapy (AC) can cause dose-related cardiomyocyte injury and death, possibly leading to left ventricular dysfunction. The most commonly accepted pathophysiological mechanism of anthracycline-induced cardiotoxicity is the oxidative stress hypothesis, which suggests that the generation of reactive oxygen species and lipid peroxidation of the cell membrane damage cardiomyocytes. However, there is considerable variability among patients in their susceptibility to anthracyclines: while many tolerate standard-dose anthracyclines without long-term complications, treatment-related cardiotoxicity may occur as early as after the first dose in other patients.

An increase in cancer survival, along with better awareness of the possible late effects of cardiotoxicity, has led to growing recognition of the need for surveillance of anthracycline-treated cancer survivors to prevent the development of heart failure.

Strategies for screening and detection of cardiotoxicity include cardiac imaging [echocardiography, nuclear imaging, cardiac magnetic resonance (CMR)] and biomarkers (troponin, natriuretic peptides).

The echocardiographic clinical standards for measuring left ventricular (LV) systolic function are LV ejection fraction (LVEF) and global longitudinal strain (GLS) with the latter as a more sensitive parameter to detect mild systolic dysfunction. There is abundant documentation that left ventricular ejection fraction (LVEF) is useful to guide clinical decisions, and emerging data show the clinical value of measuring global longitudinal strain (GLS). In the past, a study investigated the role of conventional- and speckle-tracking echocardiography in a cohort of asymptomatic children after anthracycline therapy, showing that impaired left ventricular myocardial deformation and mechanical dyssynchrony may exist after anthracycline therapy despite having normal left ventricular shortening fractions.

However, both left ventricular ejection fraction (LVEF) and global longitudinal strain (GLS) depend on left ventricular (LV) afterload and do not provide information regarding the ventricle's efficiency. Recently, the use of non-invasive myocardial work (MW) was proposed to measure left ventricular systolic function in a way that incorporates afterload and has the potential to quantify left ventricular (LV) energy waste.

Noninvasive myocardial work (MW) is a robust and reproducible index of left ventricular (LV) systolic performance. It correlates with myocardial metabolism and shows less afterload dependency than left ventricular ejection fraction (LVEF) and global longitudinal strain (GLS).

Different studies have shown the potential role of myocardial work (MW) in predicting the response to cardiac resynchronisation therapy (CRT) in patients with heart failure and reduced ejection fraction (HFrEF). However, the role of myocardial work (MW) in cancer paediatric patients has not yet been fully investigated.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric oncological patients 0-18 years
* Planned start of anthracycline therapy
* Normal left ventricular systolic function according to International Guidelines before the treatment with AC

Exclusion Criteria:

* Previous anthracycline treatment, bone marrow transplantation or chest radiation
* Pre-anthracycline treatment echocardiographic evidence of:
* More than mild pericardial effusion
* More than mild mitral regurgitation
* Poor echocardiographic acoustic window

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric oncological patients between 0 and 18 years with planned anthracycline therapy
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2033-07-21 (Estimated); Study Completion 2033-07-21 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of change in myocardial work values 1 month after first Anthracycline chemotherapy treatment in predicting a decrease of the ejection fraction at 12 months | 12 months after first Anthracycline chemotherapy treatment
  Patients will be evaluated with a complete echocardiogram, registering ejection fraction (EF) and myocardial work (MW) before the start of Anthracycline chemotherapy (AC) treatment and 1 and 12 months after first AC treatment. A Receiver operating characteristic (ROC) Curve will be constructed to evaluate the sensitivity of the myocardial work (MW) change in predicting a decrease in ejection fraction (EF). Youden index will be calculated to find the optimum value of the myocardial work (MW) discriminating the decrease or not of ejection fraction (EF).
Sensitivity of change in myocardial work values 6 months after first Anthracycline chemotherapy treatment in predicting a decrease of the ejection fraction at 12 months | 12 months after first Anthracycline chemotherapy treatment
  Patients will be evaluated with a complete echocardiogram, registering ejection fraction (EF) and myocardial work (MW) before the start of Anthracycline chemotherapy (AC) treatment and 6 and 12 months after first Anthracycline chemotherapy (AC) treatment. A Receiver operating characteristic (ROC) Curve will be constructed to evaluate the sensitivity of the myocardial work (MW) change in predicting a decrease in ejection fraction (EF). Youden index will be calculated to find the optimum value of the myocardial work (MW) discriminating the decrease or not of ejection fraction (EF).

SECONDARY OUTCOMES:
Sensitivity of change in myocardial work values 1 month after first Anthracycline chemotherapy treatment combined with Troponin-I hs and NT-proBNP biomarkers in predicting a decrease of the ejection fraction at 12 months | 12 months after first Anthracycline chemotherapy treatment
  Patients will be evaluated with a complete echocardiogram, registering ejection fraction (EF) and myocardial work (MW) before the start of Anthracycline chemotherapy (AC) treatment and 1 and 12 months after first Anthracycline chemotherapy (AC) treatment. Troponin-I hs and N-terminal pro b-type natriuretic peptide (NT-proBNP) will be evaluated in blood.
  A Receiver operating characteristic (ROC) Curve will be constructed to evaluate the sensitivity of the myocardial work (MW) change combined with Troponin-I hs and NT-proBNP biomarkers in predicting a decrease in ejection fraction (EF).
Sensitivity of change in myocardial work values 6 months after first Anthracycline chemotherapy treatment combined with Troponin-I hs and NT-proBNP biomarkers in predicting a decrease of the ejection fraction at 12 months | 12 months after first Anthracycline chemotherapy treatment
  Patients will be evaluated with a complete echocardiogram, registering ejection fraction (EF) and myocardial work (MW) before the start of Anthracycline chemotherapy (AC) treatment and 1 and 12 months after first Anthracycline chemotherapy (AC) treatment. Troponin-I hs and N-terminal pro b-type natriuretic peptide (NT-proBNP) will be evaluated in blood.
  A Receiver operating characteristic (ROC) Curve will be constructed to evaluate the sensitivity of the myocardial work (MW) change combined with Troponin-I hs and NT-proBNP biomarkers in predicting a decrease in ejection fraction (EF).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Caiffa, MD, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy, Italy